CLINICAL TRIAL: NCT05874739
Title: Validating a Digital Mobility Assessment in Parkinson's Disease Using Wearable Technology - the Mobilise-D Extension Study.
Brief Title: Mobilise-D: Extension Study
Status: Recruiting | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: KU Leuven (Other); University of Kiel (Other); University Hospital Erlangen (Other); Tel-Aviv Sourasky Medical Center (Other Government); University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: 10402; MJFF-022735 (Other Grant/Funding Number: The Michael J. Fox Foundation for Parkinson's Research.); MJFF-022736 (Other Grant/Funding Number: The Michael J. Fox Foundation for Parkinson's Research.); 323855 (Other: IRAS)
Record Dates: First submitted 2023-03-29; First posted 2023-05-25 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Aging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Cohort: Control participants who are age- and gender-matched to the PD cohort
- PD Cohort: PD Patients who have completed their participation in the Mobilise-D Clinical Validation Study

SUMMARY:
The goal of this observational study is to investigate the ability of a mobility monitor to measure and predict outcomes in Parkinson's disease (PD). It is an extension of a previous study (the Mobilise-D Clinical Validation Study) and consists of an additional follow-up visit for PD participants and the recruitment of age matched control participants. The data will inform researchers about PD disease progression and normal changes in mobility associated with aging.

DETAILED DESCRIPTION:
This study is an extension to the Mobilise-D project which aims to develop a real world digital assessment of mobility. This Extension Study will build on the work of the Clinical Validation Study (CVS) to extend the follow-up period of the Parkinson's disease (PD) cohort and to recruit an age matched control cohort. The additional data will for allow for modelling of disease progression in PD over a longer time period and inform on progression in normal ageing.

The Mobilise-D Extension Study is an observational cohort study taking place at five clinical sites across four different countries. The study will recruit up to 411 PD participants from the CVS PD cohort and 240 age and gender matched control participants.

The PD participants will attend a single follow-up visit 36 months after their initial CVS baseline visit. The control participants will attend a baseline visit and a 12-month follow-up visit. All study visits consist of the collection of descriptive, clinical, physical, neuropsychological data. Following each visit, participants are required to wear a body worn sensor for seven days continual monitoring.

A small sample of participants will be invited to take part in a semi-structured interview (Qualitative Sub Study) to better understand participants' experiences of PD symptoms and the impact they have on mobility. The investigators also want to know if the aspects of mobility that are being measured are relevant to people with PD. These interviews will take place face to face or remotely, depending on preference.

ELIGIBILITY:
Control Cohort:

Inclusion Criteria:

* Aged 50 years or over
* Able to walk 4 meters independently without walking aids
* Anticipated availability for 12 months.
* Ability to consent and comply with any study specific procedures.
* Willingness to wear a wearable sensor for mobility monitoring
* Able to read and write in first language in the respective country

Exclusion Criteria:

* Occurrence of any of the following within 3 months prior to informed consent: myocardial infarction, hospitalization for unstable angina, stroke, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), implantation of a cardiac resynchronization therapy device (CRTD), active treatment for cancer or other malignant disease, uncontrolled congestive heart disease (NYHA class >3), acute psychosis or major psychiatric disorders or continued substance abuse, other neurological or orthopaedic impairment that significantly impacts on gait
* Patients with a clinical diagnosis of PD, COPD, proximal hip fracture or MS
* History of dementia/significant cognitive impairment, or movement disorder (including essential tremor)

PD Cohort

Inclusion Criteria:

* Participant in the Mobilise-D Clinical Validation Study (CVS) PD Cohort - see below.

CVS PD Cohort:

Inclusion criteria:

* Aged 18 or over
* Patients with the clinical diagnosis of PD according to the recent criteria of the Movement Disorder Society
* Hoehn & Yahr stage I-III

Exclusion Criteria:

* History consistent with Dementia with Lewy Bodies (DLB), atypical parkinsonian syndromes (including multiple system atrophy or progressive supranuclear palsy, diagnosed according to accepted criteria)
* Repeated strokes or stepwise progression of symptoms, leading to a diagnosis of 'vascular parkinsonism'
* Drug-induced Parkinsonism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control cohort participants will be identified through Public and Patient Networks and Engagement teams and banks of volunteers already known to clinical sites. Control individuals may also be relatives or friends of PD participants. PD cohort participants will be recruited from the Mobilise-D Clinical Validation Study.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in LLFDI in controls | 12 months
  Change in the functional component score of the Late-Life Functional Disability Index (LLFDI) in control data. This assessment has 32 items, each with a scale from 5 (no difficulty) to 1 (unable to do). Raw scores are transformed into summary scores ranging from 0 (low level in ability) to 100 (high level of ability).
Change in LLFDI in PD | 36 months
  Change in the functional component score of the Late-Life Functional Disability Index (LLFDI) in PD data. This assessment has 32 items, each with a scale from 5 (no difficulty) to 1 (unable to do). Raw scores are transformed into summary scores ranging from 0 (low level in ability) to 100 (high level of ability).
Change in fall frequency in PD | 36 months
  Change in fall frequency (in previous 6 months) in PD data

SECONDARY OUTCOMES:
Difference in Real Walking Speed | 36 months (PD) and 12 months (control)
  Assess difference in Real Walking Speed between PD and control data as measured using a body worn sensor during a 7-day digital mobility assessment (DMA)
Fall frequency in controls | 12 months
  Change in fall frequency (in previous 6 months) in control data
Ability of Real Walking Speed to detect change in PD severity | 36 months
  Ability of Real Walking Speed (measured through digital mobility assessment) to detect change in PD disease severity as measured by the MDS Unified Parkinson's Disease Rating Scale (UPDRS). This assessment has 32 items, each with a scale from 5 (no difficulty) to 1 (unable to do). Raw scores are transformed into summary scores ranging from 0 (low level in ability) to 100 (high level of ability).
Ability of Real Walking Speed to predict change in physical capacity | 36 months (PD) and 12 months (control)
  Ability of Real Walking Speed (measured through digital mobility assessment) to detect change in physical capacity in PD and control data, as measured through the Late-Life Functional Disability Index (LLFDI). This assessment has 32 items, each with a scale from 5 (no difficulty) to 1 (unable to do). Raw scores are transformed into summary scores ranging from 0 (low level in ability) to 100 (high level of ability).
Ability of Real Walking Speed to predict change in PD severity | 36 months
  Ability of Real Walking Speed (measured through digital mobility assessment) to predict change in PD disease severity as measured by the MDS Unified Parkinson's Disease Rating Scale (UPDRS). This assessment has 32 items, each with a scale from 5 (no difficulty) to 1 (unable to do). Raw scores are transformed into summary scores ranging from 0 (low level in ability) to 100 (high level of ability).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Yarnall, PhD, Principal Investigator — Newcastle University
Locations (1):
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full anonymised dataset will be made available on the Mobilise-D platform
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: The dataset will be made available to the wider research community for secondary research purposes. Data may also be shared with The Michael J. Fox Foundation for Parkinson's Research (the study funder)